CLINICAL TRIAL: NCT04907760
Title: Personalized Follow-up Program in the Type 2 Diabetes Prevention
Acronym: PROXIPART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-A00375-36
Record Dates: First submitted 2021-05-25; First posted 2021-06-01 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Type2 Diabetes
Keywords: Diabetes; Metabolic Diseases; Endocrine System Diseases; Prevention
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Diseases; Endocrine System Diseases

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, randomized, controlled, two arms, multicentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With a personalized care program (Experimental): The strategy implemented is a personalized care pathway that includes participant follow-up by a nurse for 5 years with contact every 4 months for the first year, then every 6 months
  Interventions: Other: Personalized care program
- Without a personalized care program (No Intervention): The comparison strategy does not include any specific management. The patient will not receive individualized management with the nurse coordinator.

INTERVENTIONS:
Other: Personalized care program — It includes the participant follow-up by a nurse during 5 years with a contact every 4 months for the first year, then after every 6 months
  Arms: With a personalized care program

SUMMARY:
In France, the global prevalence of diabetes was estimated to 5% of the population in 2016, the type two diabetes (DT2) corresponding to 90% of cases. This number is widely underestimated because most people are untreated and undiagnosed. Due to the silent character of this disease, it is estimated that 20 à 30 % of diabetic adults have not yet been diagnosed. The conclusions, presented during the annual meeting of EASD in 2019, suggest that the precursor signs of this disease could be present until 20 years before the diagnosis.

Diabetes is a metabolic disease and people are diagnosed, in general, around 40-50 years old. The main risk factor of type II diabetes is lifestyle (rich diet, sedentary) but there is also other factors like hyperlipidemia, high blood pressure, high fasting blood sugar, stress, smoking, heredity, family history of diabetes, or gestational diabetes. This induces an increase of obesity, itself a major risk factor for type II diabetes occurrence.

From an economical aspect, chronic pathologies (including diabetes) represent 60% of health insurance expenses, even though it concerns 35% of insured persons, i.e. 20 million of patients. The average of annual reimbursement for a type 2 diabetic patient is 4890 euros. In this context, this study is the first step of thinking about a different, coordinated care approach, based on a preventive rather than curative approach.

DETAILED DESCRIPTION:
This study includes a personalized care program, including the patient follow-up by a nurse during 5 years with a contact every 4 months for the first year, then after every 6 months. The nurse will review the patient's progress and provide advice and contact with professionals: physical activity, psychologists, dieticians, endocrinologists, etc The main objective of this study is to compare, after 5 years of follow-up, the risk factors associated with type 2 diabetes, between participants who received personalized follow-up and those who did not. The secondary objectives are to compare the occurrence of type 2 diabetes, the quality of life and the compliance to the program between participants who received personalized follow-up and those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Person with a FINDRISC score ≥ 10 points
* Person who has given his/her express written and informed consent

Exclusion Criteria:

- Person already diagnosed with a type 2 diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-10-10 (Estimated); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Risk factors for type 2 diabetes in participants | 5 years
  Finnish Diabetes Risk Score (FINDRISC score) : 8 items with a total score from 0 to 26 points with 0 (no risk factor) and 26 (highest risk factor)

SECONDARY OUTCOMES:
Diabetes diagnostic | at 5 years
  measuring fasting blood glucose
The Quality of Life | at 5 years
  WHO questionary : total score out of 100, 26 questions with 5 likert scale items
program compliance | during 5 years
  Compliance is based on all the scheduled visits, the number of visits not carried out and the time during the research will be described in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Aurelie LIETAER, MD, Principal Investigator — Clinique Aguilera-RGDS

IPD SHARING:
Plan to Share IPD: No